CLINICAL TRIAL: NCT02672098
Title: Hyperthermic Intraperitoneal Chemotherapy for Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5150302
Record Dates: First submitted 2016-01-27; First posted 2016-02-03 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIPEC (Experimental): A procedure in which the internal parts of your abdomen are bathed in a warm solution of anti-cancer medications for 90 minutes.
  Interventions: Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC); Drug: Carboplatin

INTERVENTIONS:
Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC) — Hyperthermic intraperitoneal chemotherapy (HIPEC) is a procedure in which the internal parts of the abdomen are bathed in a warm solution of anti-cancer medications for 90 minutes.
  Other Names: HIPEC
Drug: Carboplatin — Carboplatin, delivered as HIPEC, will be administered at the time of surgery. Subjects will receive a single cycle of hyperthermic intraperitoneal chemotherapy.
  a single dose of carboplatin (800 mg/m2) will be administered in normal saline via intraperitoneal hyperthermic perfusion using the closed-abdomen technique. HIPEC will be continued for 90 minutes in the hyperthermic phase (41°C-43°C).

SUMMARY:
This is a phase I prospective study with the primary objective to compare the efficacy and safety of Surgical cytoreduction (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) in treatment of recurrent ovarian, primary peritoneal or fallopian tube cancers. Eligible patients consenting to this protocol will undergo their scheduled surgical procedure. After surgical cytoreduction to a residual disease ≤ 2.5 mm, a single dose of carboplatin (800 mg/m2) will be administered in normal saline via intraperitoneal hyperthermic perfusion using the closed-abdomen. HIPEC will be continued for 90 minutes in the hyperthermic phase (41°C-43°C). At 4-6 weeks after CRS, patients will go on to receive 6 cycles of standard IV platinum-based chemotherapy. The proportion of patients who are without evidence of recurrence will be assessed at 6, 9, 12 and 18 months after the day of surgery.

DETAILED DESCRIPTION:
This is a phase I prospective study with the primary objective to compare the efficacy and safety of CRS and HIPEC. The target population for this study is patients with ovarian, primary peritoneal or fallopian tube cancers undergoing secondary CRS after the first platinum-sensitive recurrence. 'Platinum-sensitive' recurrence is defined as recurrence 6 months after the completion of the primary platinum-based chemotherapy. Carboplatin, delivered as HIPEC, will be administered at the time of surgery. Subjects will receive a single cycle of hyperthermic intraperitoneal chemotherapy. Patients will then go on to receive standard platinum-based combination doublet chemotherapy (carboplatin and paclitaxel, carboplatin and gemcitabine, or carboplatin and liposomal doxorubicin) for 6 cycles.

Eligible patients consenting to this protocol will undergo their scheduled surgical procedure. After surgical cytoreduction to a residual disease ≤ 2.5 mm, a single dose of carboplatin (800 mg/m2) will be administered in normal saline via intraperitoneal hyperthermic perfusion using the closed-abdomen technique (43). HIPEC will be continued for 90 minutes in the hyperthermic phase (41°C-43°C). At 4-6 weeks after CRS, patients will go on to receive 6 cycles of standard IV platinum-based chemotherapy. Surveillance CT Chest, abdomen and pelvis with IV and oral contrast and serum CA-125 levels will be obtained at 6, 9, 12 and 18 months after the day of surgery. Recurrence-free survival will be assessed using RECIST 1.1 guideline (version 1.1).

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years old • Patients with diagnosis of epithelial ovarian carcinoma, primary peritoneal carcinoma, or fallopian tube carcinoma that has recurred >6 months since platinum-based chemotherapy (first recurrence) and are scheduled for secondary surgical evaluation/cytoreduction • ECOG/WHO Performance score of 0 to 1
* Histologic types feature would be serous, endometrioid, clear cell, undifferentiated carcinomas, transitional cell carcinoma, or mixed epithelial carcinoma • No End organ function
* Patients must have less than or equal to 2.5 mm residual disease at the completion of the secondary surgery to be eligible for the study

Exclusion Criteria:

* Subjects who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded • Subjects with invasive malignancies or had any evidence of the other cancer present within the last 3 years
* Tumors of low malignant potential • Patients with active coronary artery disease • Patients with known acute hepatitis • Patients with restrictive or obstructive pulmonary disease
* Patient with extra-abdominal metastatic disease • Immuno-compromized patients
* Known carboplatin or Cisplatin allergy • Life expectancy < 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival compared to historical controls | 6 months after the day of surgery
  Surveillance CT Chest, abdomen and pelvis with IV and oral contrast and serum CA-125 levels will be obtained at 6 months after the day of surgery. Recurrence-free survival will be assessed using RECIST 1.1 guideline (version 1.1).
Recurrence-free survival compared to historical controls | 9 months after the day of surgery
  Surveillance CT Chest, abdomen and pelvis with IV and oral contrast and serum CA-125 levels will be obtained at 9 months after the day of surgery. Recurrence-free survival will be assessed using RECIST 1.1 guideline (version 1.1).
Recurrence-free survival compared to historical controls | 12 months after the day of surgery
  Surveillance CT Chest, abdomen and pelvis with IV and oral contrast and serum CA-125 levels will be obtained at 12 months after the day of surgery. Recurrence-free survival will be assessed using RECIST 1.1 guideline (version 1.1).
Recurrence-free survival compared to historical controls | 18 months after the day of surgery
  Surveillance CT Chest, abdomen and pelvis with IV and oral contrast and serum CA-125 levels will be obtained at 18 months after the day of surgery. Recurrence-free survival will be assessed using RECIST 1.1 guideline (version 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Mazdak Momeni, MD, Principal Investigator — Loma Linda University Cancer Center
Locations (1):
- Women's Cancer and Surgical Oncology Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- See also: Intraperitoneal Cisplatin and Paclitaxel in Ovarian Cancer — https://pubmed.ncbi.nlm.nih.gov/16394300/